CLINICAL TRIAL: NCT03745976
Title: Evaluation of a New Long-term Total Articular Prosthesis Follow-up Strategy by Simple Questionnaire and Radiography
Brief Title: Questionnaire and Radiography for Prosthesis Follow-up
Acronym: Follow-up
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-412; 2018-A01022-53 (Other: 2018-A01022-53)
Record Dates: First submitted 2018-10-19; First posted 2018-11-19 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Hip and Knee Arthroplasties; Without Known Complication; Annual Follow-up
Keywords: follow-up; total knee arthroplasty; total hip arthroplasty
MeSH Terms: interventions — Surveys and Questionnaires; X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: a new long-term total articular prosthesis follow-up strategy by simple questionnaire and radiography (questionnaire and Xray for all patients)
  Interventions: Procedure: questionnaire and Xray for all patients

INTERVENTIONS:
Procedure: questionnaire and Xray for all patients — questionnaire and Xray for all patients

SUMMARY:
Ever-evolving prosthetic activity as described in a Swedish study that predicts 469 TKA per 10,000 inhabitants in 2130. Increased consultation of controls and post-arthroplasty follow-up is expected. There is a legal obligation to ensure long-term follow-up without official recommendation on follow-up procedures. The objective is to compare a consultation + Xray by the surgeon versus an Xray and a questionnaire completed by the patient who had a knee or hip replacement. This is to demonstrate the equivalence of both.

All patients who come back for an annual check of a prosthesis should complete this questionnaire and perform an X-ray of their prosthesis. The study lasts one year and includes all the patients with a previous knee or hip arthroplasty.

The result of the questionnaire and Xray will be compared to that of the consultation and Xray.

DETAILED DESCRIPTION:
An english study published an article showing that a follow up by questionnaire versus a consultation was also effective.

For this study, investigator is going to take back all the patients having to return to consultation in 2017. . Normally at 3 months, 1, 3, 5, 10, 15 and 20 years post-operatively.

Thus investigator will be able to see the number of patients seen in consultation compared to the theoretical number The purpose of this study is to highlight the non-inferiority of the questionnaire compared to the consultation for screening for complications at 10 years.

If this proves to be the case, only complicating patients could be reviewed by calling them to the radio and their questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a primary total hip or total knee arthroplasty that must be seen again in 2017. Normally at 3 months, 1 years, 3, 5, 10, 15 and 20 years post-operatively

Exclusion Criteria:

* Patients who have previous complications with their joint replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had a primary total hip or total knee arthroplasty that must be seen again in 2017
Sampling Method: Non-Probability Sample
Enrollment: 656 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Patients seen in consultation follow-up or not (yes / no). | at 3 months
  Feasibility study of a new strategy of follow-up by questionnaire
Patients seen in consultation follow-up or not (yes / no). | at 1year
  Feasibility study of a new strategy of follow-up by questionnaire
Patients seen in consultation follow-up or not (yes / no). | at 3 years
  Feasibility study of a new strategy of follow-up by questionnaire
Patients seen in consultation follow-up or not (yes / no). | at 5 years
  Feasibility study of a new strategy of follow-up by questionnaire
Patients seen in consultation follow-up or not (yes / no). | at 10 years
  Feasibility study of a new strategy of follow-up by questionnaire
Patients seen in consultation follow-up or not (yes / no). | at 15 years
  Feasibility study of a new strategy of follow-up by questionnaire
Patients seen in consultation follow-up or not (yes / no). | at 20 years
  Feasibility study of a new strategy of follow-up by questionnaire

SECONDARY OUTCOMES:
economic impact (Number of working day) | at 3 months, 1, 3, 5, 10, 15 and 20 years post-operatively.
  Number of working day in days
economic impact (Number of consultations) | at 3 months, 1, 3, 5, 10, 15 and 20 years post-operatively.
  Number of consultations with the surgeon,
economic impact (Number of radiography) | at 3 months, 1, 3, 5, 10, 15 and 20 years post-operatively.
  Number of radiography realized by the patient
economic impact (Cost phone call) | at 3 months, 1, 3, 5, 10, 15 and 20 years post-operatively.
  According to the number of realized phone call
Evaluation of the feasibility of the questionnaire for detection of certain complications | at 3 months, 1, 3, 5, 10, 15 and 20 years post-operatively.
  Evaluation of the feasibility of the questionnaire method

CONTACTS AND LOCATIONS:
Overall Officials: Roger ERIVAN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France